CLINICAL TRIAL: NCT04081272
Title: Effect of Glucose-6-phosphate Dehydrogenase Deficiency on Donor Red Blood Cell Storage
Brief Title: Effect of G6PD Deficiency on Red Blood Cell Storage
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: New York Blood Center (Other)
Responsible Party: Sponsor
Other Study IDs: AAAJ6862
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: G6PD Deficiency
Keywords: transfusion; post-transfusion recovery
MeSH Terms: conditions — Glucosephosphate Dehydrogenase Deficiency | interventions — sodium chromate(VI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected to conduct a complete blood count (CBC), testing for the presence of abnormal hemoglobin types (hemoglobinopathy screen), blood type and antibody screen, and confirmation of G6PD deficiency by measuring enzyme activity. In addition, DNA will be extracted and preserved for genetic testing for G6PD deficiency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- G6PD-normal: Donated blood from G6PD-normal subjects
  Interventions: Drug: Sodium Chromate Cr51
- G6PD-deficient: Donated blood from G6PD-deficient subjects
  Interventions: Drug: Sodium Chromate Cr51

INTERVENTIONS:
Drug: Sodium Chromate Cr51 — Sodium Chromate Cr 51 will be used to perform a red blood cell recovered study 24 hours post-transfusion.
  Other Names: Chromitope

SUMMARY:
The proposed study will determine whether G6PD-deficient RBCs store differently than normal RBCs under standard blood banking conditions. The investigators plan to screen a large number of healthy male volunteers for G6PD deficiency in order to identify 10 G6PD deficient and 30 matched normal individuals using a blood sample obtained from a finger-stick. The identified individuals will then be asked to donate a unit of blood that will be stored for up to 42 days and various tests will be performed on these units during storage. At 6 weeks of storage a portion of the unit will be radioactively labeled and re-infused into the volunteer. Blood samples will be drawn before, during, and after the infusion to measure how well or poorly the red blood cells survive after transfusion.

DETAILED DESCRIPTION:
Glucose-6-phosphate dehydrogenase (G6PD) deficiency is the most common enzyme deficiency, affecting approximately 400 million people world-wide. It manifests as red blood cell (RBC) destruction in response to oxidative stress, which can be precipitated by infection, and by the ingestion of certain medications and foods. The prevalence of G6PD deficiency varies among populations and is most commonly found in individuals from sub-Saharan Africa, the Mediterranean region, and south-east Asia. Although in most studies G6PD-deficient individuals have normal RBC survival at steady-state, this may vary based upon the G6PD variant present, and some individuals may have shortened RBC survival. While it is not routine practice to screen blood donors for G6PD deficiency, G6PD deficient donor RBCs may store more poorly than normal RBCs. In addition, the transfusion of stored G6PD-deficient RBCs may result in decreased RBC survival after transfusion compared to RBCs from normal donors.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Weight greater than 110 pounds
* Hemoglobin greater than 11.5 g/dL
* African (e.g., Afro-American, Afro-Caribbean, Sub-Saharan), Asian, Hispanic, Middle Eastern, or Mediterranean (e.g., Italian, Greek) based on mother's ancestry
* English speaking

Exclusion Criteria:

* Presence of hemoglobin variant
* Ineligible for donation based on the New York Blood Center donor autologous questionnaire
* Systolic blood pressure >180 or <90 mm Hg, diastolic blood pressure >100 or <50 mm Hg
* Heart rate <50 or >100
* Temperature >99.5°F prior to donation
* Temperature >100.4°F or subjective feeling of illness prior to transfusion (this criterion is to avoid concurrent illness affecting post-transfusion measurements)
* Positive results on standard blood donor infectious disease testing

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male volunteers will be screened for G6PD deficiency in order to identify 10 G6PD deficient and 30 matched normal individuals using a blood sample obtained from a finger-stick.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
24-hour post-transfusion red blood cell recovery | 24 hours
  Percentage of radio-labeled red blood cells remaining 24 hours after infusion

SECONDARY OUTCOMES:
In vitro hemolysis rate | 42 days
  Percent hemolysis in the red blood cell unit in vitro

OTHER OUTCOMES:
Number of samples with metabolites detected | Pre-donation to 42 days after donation
  Metabolomics analysis: metabolites that are representative of major metabolic pathways will be measured in the red blood cells or supernatant during storage. Quantitative measurements will be performed using high performance liquid chromatography and mass spectrometry and the data obtained will be analyzed to detect correlations with the primary outcome measure of 24-hour post-transfusion red blood cell recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Richard O Francis, MD, PhD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - New York Blood Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
We will share all individual study data results upon request once the study is published.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: upon request once the study is published
Access Criteria: email study PI to request data

REFERENCES:
- [Derived] Francis RO, D'Alessandro A, Eisenberger A, Soffing M, Yeh R, Coronel E, Sheikh A, Rapido F, La Carpia F, Reisz JA, Gehrke S, Nemkov T, Thomas T, Schwartz J, Divgi C, Kessler D, Shaz BH, Ginzburg Y, Zimring JC, Spitalnik SL, Hod EA. Donor glucose-6-phosphate dehydrogenase deficiency decreases blood quality for transfusion. J Clin Invest. 2020 May 1;130(5):2270-2285. doi: 10.1172/JCI133530. PMID 31961822